CLINICAL TRIAL: NCT06274658
Title: The Effects of an Acute High-intensity Interval Training on Heart and Brain Function in People With Spinal Cord Injury
Brief Title: The Effects of an Acute High-intensity Exercise on Heart and Brain Function in People With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Wenjie Ji, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00006517
Record Dates: First submitted 2024-02-13; First posted 2024-02-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Autonomic Nervous System Disease; Spinal Cord Injuries; Cognition
MeSH Terms: conditions — Spinal Cord Injuries | interventions — High-Intensity Interval Training

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Spinal Cord Injury: This group includes people with spinal cord injury and the level of injury is at the 6th thoracic vertebra or above.
  Interventions: Behavioral: High-intensity interval exercise
- Non-injured Controls: This group includes age- and sex-matched non-injured control participants.
  Interventions: Behavioral: High-intensity interval exercise

INTERVENTIONS:
Behavioral: High-intensity interval exercise — Three high-intensity exercise bouts, each at 100% of maximal power output for 20 seconds, interspersed with active recovery periods of 120 seconds at 10% of maximal power output.

SUMMARY:
The heart and brain are regulated by the autonomic nervous system. Control of these organs can be disrupted in people with spinal cord injury (SCI). This may affect their ability to regulate blood pressure during daily activities and process the high-level information. Previous studies show that high-intensity exercise induces better outcomes on heart and information processing ability in non-injured people compared to moderate-intensity exercise. However, it is unknown the effects of high-intensity exercise on heart and brain function in people with SCI. Therefore, this study aims to examine the effects of a single bout of high-intensity interval training on heart and brain function in this people with SCI compared to age- and sex-matched non-injured controls.

DETAILED DESCRIPTION:
This study will be a cohort control study involving two groups: individuals with SCI, whose level of injury is at the 6th thoracic vertebra or above, and age- and sex-matched controls. Eligible participants will be asked to visit the Laboratory located at 115 Kimball Tower, University at Buffalo South Campus, twice. The first visit takes up to 3 hours, and the second visit takes up to 5 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with a traumatic or non-traumatic spinal cord injury and have ≥4/5 strength in at least one cervical 5 myotome (elbow flexors), allowing to utilize the arm ergometer and level of injury at or above the 6th thoracic vertebra
2. Classified as A, B, C, D (motor and sensory complete or incomplete) on the American Spinal Injury Association (ASIA) Impairment Scale (AIS)
3. Longer than 6 months post the onset of injury and have been discharged to the community from inpatient rehabilitation prior to enrollment
4. English is the first language
5. At least one of the cerebral arteries (i.e., middle cerebral artery and/or posterior cerebral artery) can be found via transcranial Doppler

Exclusion Criteria:

1. Medical conditions that preclude exercise, such as unstable angina, uncontrolled arrhythmias, a recent history of congestive heart failure that has not been evaluated and effectively treated, severe valvular disease, uncontrolled hypertension (i.e., resting systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 105 mmHg)
2. Moderate-severe traumatic brain injury
3. Diabetes
4. Color blindness
5. Pre-existing shoulder injuries
6. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include people with SCI with level of injury T6 or above and age- and sex-matched non-injured controls.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Low frequency of systolic blood pressure variability | Baseline, Physiological tests pre- and 10 minutes post-exercise
  Biomarker for autonomic nervous system function
High frequency of heart rate variability | Baseline, Physiological tests pre- and 10 minutes post-exercise
  Biomarker for autonomic nervous system function
Blood pressure | Baseline, Physiological tests pre- and 10 minutes post-exercise
  Biomarker for autonomic nervous system function
Heart rate | Baseline, Physiological tests pre- and 10 minutes post-exercise
  Biomarker for autonomic nervous system function

SECONDARY OUTCOMES:
Cerebral blood flow velocity | Baseline, cognitive tests pre- and 10-minutes post-exercise
  Biomarker for cerebrovascular function
Symbol Digit Matched Test score | Baseline, cognitive tests pre- and 10-minutes post-exercise
  Assessment for cognitive function
California Verbal Learning Test score | Baseline, cognitive tests pre- and 10-minutes post-exercise
  Assessment for cognitive function
Color-Word Stroop Test score | Baseline, cognitive tests pre- and 10-minutes post-exercise
  Assessment for cognitive function
Controlled Word Association Task score | Baseline, cognitive tests pre- and 10-minutes post-exercise
  Assessment for cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Ji, MS, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, South Campus, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ji W, Wecht JM, Jo HJ, Stefanovic F, Miecznikowski J, Chiaravalloti ND, Sisto SA. Effects of a single bout of high-intensity-interval exercise on cardiovascular autonomic, cerebrovascular, and cognitive function in people with spinal cord injury: A study protocol. PLoS One. 2025 Jul 1;20(7):e0326861. doi: 10.1371/journal.pone.0326861. eCollection 2025. PMID 40591703